CLINICAL TRIAL: NCT01256567
Title: A Phase 1b Study of Docetaxel in Combination With Ramucirumab (IMC-1121B) Drug Product in Patients With Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of Ramucirumab (IMC-1121B) in Participants With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14200; CP12-1028 (Other: ImClone Systems); I4T-IE-JVBX (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ramucirumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ramucirumab and docetaxel combination (Experimental)
  Interventions: Biological: Ramucirumab; Drug: Docetaxel

INTERVENTIONS:
Biological: Ramucirumab — Ramucirumab administered as an intravenous (I.V.) infusion at a dose of 10 milligrams per kilogram (mg/kg) every 3 weeks.
  Other Names: IMC-1121B; LY3009806
Drug: Docetaxel — Docetaxel administered by intravenous (I.V.) infusion at a dose of 75 milligrams per square meter (mg/m^2) every 3 weeks.

SUMMARY:
The primary objective of this study is to investigate the safety and tolerability of the anti-VEGFR-2 monoclonal antibody ramucirumab drug product in combination with docetaxel in Japanese participants with metastatic, or locally advanced breast cancer, with the aim of confirming the recommended dose of ramucirumab drug product (DP) in combination with docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* The participant is Japanese
* The participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* The participant has a histopathologically or cytologically confirmed diagnosis of breast adenocarcinoma that is now metastatic or locally-recurrent and inoperable with curative intent
* The participant has measurable and/or non-measurable disease
* The participants' primary and/or metastatic tumor is Human Epidermal Growth Factor Receptor 2 (HER2) negative
* The participant received neo adjuvant or adjuvant taxane therapy ≥ 6 months prior to the study
* The participant received neo adjuvant or adjuvant biologic therapy ≥ 6 weeks prior to the study
* The participant completed all prior radiotherapy ≥ 3 weeks prior to the study registration date
* The participant received prior hormonal therapy for breast cancer in the neo adjuvant, adjuvant,and/or the metastatic setting ≥ 2 weeks prior to the study registration date
* The participant's left ventricular ejection fraction (LVEF) is within normal ranges
* The participant has adequate hematologic, hepatic, and coagulation function.
* Eligible participants of reproductive potential agree to use adequate contraceptive methods (hormonal or barrier methods) during the study period and for 12 weeks after the last dose of study medication

Exclusion Criteria:

* The participant has a concurrent active malignancy other than breast adenocarcinoma, adequately treated non-melanomatous skin cancer, or other non-invasive carcinoma or in situ neoplasm. Participants with previous treatment of malignancy is eligible, provided that she has been disease free for >3 years
* The participant has a known sensitivity to docetaxel
* The participant has a known sensitivity to agents of similar biologic composition as ramucirumab
* The participant has a history of chronic diarrheal disease within 6 months prior to the study registration date
* The participant has received irradiation to a major bone marrow area within 30 days prior to the study registration date
* The participant has received any experimental agents within 4 weeks prior to the study registration date
* The participant has a history of uncontrolled hereditary or acquired bleeding or thrombotic disorders
* The participant has Grade 3-4 bleeding within 3 months prior to the study registration date
* The participant has an ongoing or active infection requiring antibiotic, antifungal, or antiviral therapy
* The participant has uncontrolled hypertension, symptomatic congestive heart failure, psychiatric illness, or any other serious uncontrolled medical disorders
* The participant has brain metastases
* The participant has known human immunodeficiency virus infection or acquired immunodeficiency syndrome related illness
* The participant is pregnant or lactating
* The participant has not fully recovered from effects of prior chemotherapy
* The participant has undergone major surgery within 28 days prior to the study registration date

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- Japan (4):
  - ImClone Investigational Site, Hidaka
  - ImClone Investigational Site, Matsuyama
  - Imclone Investigational Site, Nagoya
  - ImClone Investigational Site, Osaka

RESULTS

PARTICIPANT FLOW:
Groups:
- Ramucirumab and Docetaxel Combination: Docetaxel: Docetaxel administered by intravenous infusion at a dose of 75 milligrams per square meter (mg/m^2) every 3 weeks.
  Ramucirumab: Ramucirumab (IMC-1121B) administered as an intravenous infusion at a dose of 10 milligrams per kilogram (mg/kg) every 3 weeks.
Period: Overall Study
Arm/Group | Ramucirumab and Docetaxel Combination
Started | 7
Received at Least 1 Dose of Study Drug | 7
Completed | 6
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Ramucirumab and Docetaxel Combination: Docetaxel: Docetaxel administered by intravenous infusion at a dose of 75 milligrams per square meter (mg/m^2) every 3 weeks.
  Ramucirumab: Ramucirumab administered as an intravenous infusion at a dose of 10 milligrams per kilogram (mg/kg) every 3 weeks.
Arm/Group | Ramucirumab and Docetaxel Combination
Number analyzed (Participants) | 7
Age, Customized [Number; unit: participants]
  Between 20 and 65 years | 6
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 7
  American Indian or Alaska Native | 0
  Black or African American | 0
  Native Hawaiian or Other Pacific Islander | 0
  White | 0
  Other | 0
Region of Enrollment [Number; unit: participants]
  Japan | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number participants with drug related dose-limiting toxicities (DLT) during Cycle 1; ramucirumab related: treatment-emergent adverse events (TEAE), serious adverse events (SAE), Grade 3 or higher TEAE, or TEAE leading to discontinuation or ramucirumab dose modification. DLT=G4 neutropenia >7days; G ≥3 neutropenia with fever ≥38.5°C requiring IV antibiotics or bacteriemia or sepsis; G4 thrombocytopenia; G ≥3 thrombocytopenia with bleeding requiring platelets; G≥3 prothrombin time and/or partial thromboplastin time in absence of anticoagulants; G≥2 hyperbilirubinemia ≥5 days; QTc >500 milliseconds (ms) or increase ≥100 ms or arrhythmia; G≥4 or uncontrollable hypertension; G≥3 nonhematologic toxicity (excluding G3: hypersensitivity, injection-site reaction, arthralgia/myalgia, asthenia/fatigue, diarrhea without loperamide therapy, nausea/vomiting without antiemetics, transient G3/4 elevation of aminotransferases); treatment delay >2 weeks due to toxicity.
Time Frame: Baseline up to data cut off (approximately 48.3 weeks)
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ramucirumab and Docetaxel Combination
Number analyzed (Participants) | 7
participants
  Dose Limiting Toxicity (DLT) during Cycle 1 | 2
  TEAE related to ramucirumab | 7
  SAE related to ramucirumab | 4
  TEAE of Grade ≥3 related to ramucirumab | 6
  TEAE resulting in ramucirumab discontinuation | 3
  TEAE with ramucirumab dose modification/delay | 5

2. Secondary Outcome: Serum Anti-IMC-1121B Antibody Assessment (Immunogenicity)
Description: The number of participants with a positive anti-IMC-1121B titer at any point during the study.
Time Frame: Baseline up to data cut off (approximately 48.3 weeks)
Population: All participants with evaluable antibody assessment data.
Measure: Number; unit: participants
Arm/Group | Ramucirumab and Docetaxel Combination
Number analyzed (Participants) | 7
participants | 0

3. Secondary Outcome: Maximum Concentration (Cmax) of Ramucirumab
Description: Cmax (Cycle 1) and Cmax at steady state (Cmax,ss, Cycle 4) of ramucirumab are provided.
Time Frame: Day 1 of Cycle 1 and Cycle 4 (cycle=21 days)
Population: All participants with evaluable Cmax data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Ramucirumab and Docetaxel Combination
Number analyzed (Participants) | 7
micrograms per milliliter (mcg/mL)
  Cmax at Cycle 1 | 261 (22)
  Cmax,ss at Cycle 4 (n=6) | 335 (22)

4. Secondary Outcome: Area Under the Curve (AUC) of Ramucirumab
Description: AUC from time zero to infinity (AUC[0-inf], Cycle 1) and at steady state (AUC tau, Cycle 4) of ramucirumab are provided.
Time Frame: Day 1 of Cycles 1 and 4 (cycle=21 days)
Population: All participants with evaluable AUC data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*day/milliliter (mcg*day/mL)
Arm/Group | Ramucirumab and Docetaxel Combination
Number analyzed (Participants) | 7
micrograms*day/milliliter (mcg*day/mL)
  AUC(0-inf) at Cycle 1 | 1700 (25)
  AUC tau at Cycle 4 (n=6) | 2320 (24)

5. Secondary Outcome: Half Life (t 1/2) of Ramucirumab
Time Frame: Day 1 of Cycles 1 and 4 (cycle=21 days)
Population: All participants with evaluable t1/2 data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Ramucirumab and Docetaxel Combination
Number analyzed (Participants) | 7
days
  t1/2 at Cycle 1 | 6.57 (49)
  t1/2 at Cycle 4 (n=6) | 11.9 (26)

6. Secondary Outcome: Clearance (Cl) of Ramucirumab
Description: Clearance (Cycle 1) and at steady state (Clss, Cycle 4) of ramucirumab are provided.
Time Frame: Day 1 of Cycle 1 and Cycle 4 (cycle=21 days)
Population: All participants with evaluable clearance data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per hour (mL/hr)
Groups:
- Ramucirumab and Docetaxel Combination: Docetaxel : Docetaxel administered by intravenous infusion at a dose of 75 milligrams per square meter (mg/m^2) every 3 weeks.
  Ramucirumab : Ramucirumab administered as an intravenous infusion at a dose of 10 milligrams per kilogram (mg/kg) every 3 weeks.
Arm/Group | Ramucirumab and Docetaxel Combination
Number analyzed (Participants) | 7
milliliters per hour (mL/hr)
  Clearance at Cycle 1 | 13.6 (24)
  Clearance at steady state (Clss) at Cycle 4 (n=6) | 10.2 (24)

7. Secondary Outcome: Steady State Volume of Distribution (Vss) of Ramucirumab
Time Frame: Day 1 of Cycle 1 and 4 (cycle=21 days)
Population: All participants with evaluable Vss data at the specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)
Arm/Group | Ramucirumab and Docetaxel Combination
Number analyzed (Participants) | 7
liters (L)
  Vss at Cycle 1 | 2.96 (32)
  Vss at Cycle 4 (n=6) | 3.92 (18)

ADVERSE EVENTS:
Arm/Group | Ramucirumab and Docetaxel Combination
Serious Adverse Events (participants affected / at risk) | 7/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab and Docetaxel Combination (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Cardiac failure (Cardiac disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab and Docetaxel Combination (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (9)
Palpitations (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Asthenopia (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (2)
Lacrimation increased (Eye disorders) | 3 (3)
Myodesopsia (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (6)
Diarrhoea (Gastrointestinal disorders) | 2 (4)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 2 (8)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3)
Periodontitis (Gastrointestinal disorders) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 3 (9)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest discomfort (General disorders) | 1 (2)
Face oedema (General disorders) | 4 (6)
Fatigue (General disorders) | 2 (4)
Infusion related reaction (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Malaise (General disorders) | 4 (19)
Mucosal inflammation (General disorders) | 4 (9)
Oedema peripheral (General disorders) | 7 (16)
Pyrexia (General disorders) | 2 (3)
Cystitis (Infections and infestations) | 1 (4)
Nasopharyngitis (Infections and infestations) | 5 (8)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Blood urine (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 5 (17)
Platelet count decreased (Investigations) | 1 (4)
Platelet count increased (Investigations) | 1 (2)
Weight increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (2)
White blood cell count increased (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (10)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dysgeusia (Nervous system disorders) | 4 (10)
Headache (Nervous system disorders) | 2 (3)
Lacunar infarction (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (5)
Presyncope (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (5)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (12)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkeratosis palmaris and plantaris (Skin and subcutaneous tissue disorders) | 1 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 5 (5)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (5)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.